CLINICAL TRIAL: NCT01963910
Title: Double-blind Trial of Mannitol Cream to Block the Effect of Capsaicin Cream
Acronym: LipTRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Helene Bertrand, Clinical instructor Department of Family Practice, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H13-01551
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Pain
Keywords: Mannitol; TRPV1 receptor; Pain; Burning pain; neuropathy; neuropathic pain
MeSH Terms: conditions — Pain; Neuralgia | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol in vehicle cream (Active Comparator): Once the capsaicin has been removed, .2 mL of 30% mannitol in vehicle cream will be applied to one half of the upper lip and kept there for 10 minutes.
  Interventions: Drug: 30% Mannitol in vehicle cream
- Vehicle Cream (Placebo Comparator): Once the capsaicin has been removed, .2 mL of vehicle cream will be applied to the other half of the upper lip and kept there for 10 minutes.
  Interventions: Drug: vehicle cream

INTERVENTIONS:
Drug: 30% Mannitol in vehicle cream — applied to one half of the upper lip following removal of capsaicin cream.
  Other Names: mannitol cream; Mannitol; mannite; manna sugar; C6H8(OH)6
  Arms: Mannitol in vehicle cream
Drug: vehicle cream — application to the other half of the upper lip following capsaicin cream removal
  Arms: Vehicle Cream

SUMMARY:
Capsaicin is a TRPV1 (transient receptor potential vanilloid 1) agonist, causing pain upon application. The investigators wish to determine whether mannitol blocks the effect of capsaicin application. As both cream bases are identical and mannitol addition is the only difference between the creams, if the mannitol cream is more effective in blocking the effect of capsaicin on the TRPV1 (transient receptor potential vanilloid 1) receptor, the investigators will have established that mannitol down-regulates or blocks the TRPV1 (transient receptor potential vanilloid 1) receptor.

DETAILED DESCRIPTION:
Capsaicin cream, which stimulates the TRPV1 (transient receptor potential vanilloid 1) receptor, causing a burning sensation, will be applied to both halves of the upper lip until a burning sensation with 8/10 intensity on an NRS (Visual Analog Scale) scale is experienced or five minutes have elapsed. Following this, the capsaicin cream will be wiped off and 30% mannitol in vehicle cream ( isopropyl palmitate, caprylic capric triglyceride, propylene glycol, ceteareth 20, cetearyl alcohol, glyceryl stearate, polyethylene glycol 100 stearate, dimethicone, octyldodecanol, lecithin, ethylhexyl glycerin and phenoxy ethanol) will be applied to one half of the upper lip, and vehicle cream alone will be applied to the other half. Cream assignment will be randomized and neither the subject nor the person applying the cream will know which half upper lip has which cream. Every minute for 10 minutes, the heat sensation felt in each half upper lip will be measured, using a visual scale from 0 to 10. A repeated measures analysis of variance will compare the NRS (Visual Analog Scale) scores from the 30% mannitol cream, to the NRS (Visual Analog Scale)scores from the vehicle cream. Significance will be accepted if P less than .05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 80 years

Exclusion Criteria:

* Diet containing capsaicin (Cayenne pepper, capsicum) (spicy foods), more than once a week.
* Meal containing capsaicin (spicy foods) within 5 days prior to the experiment.
* Any lesion, cracking, cold sore or abrasion on the lips
* Inability to tolerate capsaicin containing "spicy foods"
* Wearing lipstick or lip balm on the upper lip
* Inability to fill out an NRS pain scale
* Use of painkilling medication, within 24 hours of the study.
* Allergy to any of the ingredients of the creams, or to mannitol
* History of contact or allergic dermatitis
* Pregnant or nursing women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
NRS heat score, once per minute | 15 minutes per subject
  Every minute after capsaicin cream application, subject will indicate NRS (numerical rating scale)heat score. When the score has reached 8/10 or after five minutes, the cream will be removed. The time needed to reach 8/10 heat score and the heat score achieved, or the score at five minutes will be recorded. Following application of the test creams, NRS (Visual Analog Scale) heat scores will be recorded once per minute for each side for 10 minutes.

SECONDARY OUTCOMES:
Side effects of capsaicin cream on upper lip | One hour
  The subject will be observed for redness, swelling, or other side effects following the capsaicin cream application. These side effects will be recorded

OTHER OUTCOMES:
Side effects of test creams | one hour
  The subjects will be observed for side effects of the mannitol cream or the vehicle cream

CONTACTS AND LOCATIONS:
Overall Officials: Helene Bertrand, MD, CM, CCFP, Principal Investigator — Department of family practice, University of British Columbia
Locations (1):
- Dr. Helene Bertrand Inc., 220-1940 Lonsdale Ave., North Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Ngom PI, Dubray C, Woda A, Dallel R. A human oral capsaicin pain model to assess topical anesthetic-analgesic drugs. Neurosci Lett. 2001 Dec 28;316(3):149-52. doi: 10.1016/s0304-3940(01)02401-6. PMID 11744224
- [Background] Boudreau SA, Wang K, Svensson P, Sessle BJ, Arendt-Nielsen L. Vascular and psychophysical effects of topical capsaicin application to orofacial tissues. J Orofac Pain. 2009 Summer;23(3):253-64. PMID 19639105
- [Derived] Bertrand H, Kyriazis M, Reeves KD, Lyftogt J, Rabago D. Topical Mannitol Reduces Capsaicin-Induced Pain: Results of a Pilot-Level, Double-Blind, Randomized Controlled Trial. PM R. 2015 Nov;7(11):1111-1117. doi: 10.1016/j.pmrj.2015.05.002. Epub 2015 May 12. PMID 25978942